CLINICAL TRIAL: NCT04802460
Title: Virtual Reality Effects on Acute Pain During Office Hysteroscopy: A Randomized Control Study
Brief Title: Virtual Reality Effects on Pain During Hysteroscopy Hysteroscopy: A Randomized Control Trial
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001687
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Pain and Hysteroscopy
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): Patients assigned to the VR group will be engaged with the VR using a publicly available VR set. Both study groups will be directed to take 800mg ibuprofen 1 hour prior to scheduled surgery as standard pain management in our office.
  Interventions: Device: Virtual reality headset (The Guided Meditation VR App through Oculus Go headset)
- control arm (No Intervention): Patients in the control arm will undergo standard of care office hysteroscopy. Both study groups will be directed to take 800mg ibuprofen 1 hour prior to scheduled surgery as standard pain management in our office.

INTERVENTIONS:
Device: Virtual reality headset (The Guided Meditation VR App through Oculus Go headset) — Patients assigned to the VR condition will engage with the VR using The Guided Meditation VR App through Oculus Go headset. They will enjoy up to a 10 minute video of an environment of their choosing. During this video they will listen to calming music and a guided meditation session.
  Arms: virtual reality

SUMMARY:
The Objective of this study is to compare pain levels in women undergoing office-based hysteroscopies using Virtual Reality versus control in a randomized control prospective trial.

DETAILED DESCRIPTION:
The primary aim of this study is to see if virtual reality can decrease pain intensity during office hysteroscopies using a 100mm Visual Analogue Scale (VAS).

A secondary aim will be to monitor heart rate for patients using virtual reality versus the controls during the procedure. Another secondary aim will be to time the length of the procedure as it is possible if pain perception is reduced, the procedure can be completed faster. Lastly, we would also want to evaluate both patient and surgeon satisfaction of the procedure with or without virtual reality by using a satisfaction questionnaire to assess for patients satisfaction with the procedure, with the VR intervention, perceived realism of VR game, and measure simulator sickness related to the VR game.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be women over the age of 18 presenting for office hysteroscopy.

Exclusion Criteria:

Exclusion criteria included patients with visual or auditory impairment that would interfere with their ability to use the virtual reality set, English language non-fluency, history of opioid dependence/abuse, current narcotic use, or desire for narcotic use during the procedure.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
pain scale | 10 minutes
  The primary aim of this study is to see if virtual reality can decrease pain intensity during office hysteroscopies using a 100mm Visual Analogue Scale (VAS).

SECONDARY OUTCOMES:
heart rate changes | 10 minutes
  The secondary outcomes will be change in pain score and change in participant's HR throughout the procedure to assess for sympathetic evidence of pain and anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- MHRI IRB, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No